CLINICAL TRIAL: NCT00997789
Title: Bioequivalence Evaluation of Two Rebamipide Preparations After a Single Oral Dose to Healthy Korean Volunteers
Brief Title: Bioequivalence of Rebamipide in Korean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Institute of Bioequivalence and Bridging Study, College of Pharmacy, CNU (Unknown)
Responsible Party: Yong-Bok Lee, Professor and Director, Institute of Bioequivalence and Bridging Study, College of Pharmacy, CNU
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IBBS-BE-REBAMIPIDE-KYUNGDONG
Record Dates: First submitted 2009-10-14; First posted 2009-10-19 (Estimated); Last update posted 2009-10-19 (Estimated); Status verified 2009-10

CONDITIONS: Therapeutic Equivalency; Pharmacogenetics
Keywords: Rebamipide; Bioequivalence; ABCB1 genetic polymorphisms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rebamipide, Serum concentration, Tablet (Experimental): The test preparation, Rebamide® (containing 100 mg of rebamipide; lot No. KP005; expiration date, April 2010; Kyungdong Pharmaceutical Company, Seoul, Korea) and the reference preparation, Mucosta® (containing 100 mg of rebamipide; lot No. MC704067; expiration date, May 2010; Korea Otsuka Pharmaceuticals Co., Ltd., Seoul, Korea)
  Interventions: Drug: Rebamide

INTERVENTIONS:
Drug: Rebamide — Rebamipide 100 mg Tablet, three times a day
  Other Names: Mucosta® (Korea Otsuka Pharmaceuticals Co.)

SUMMARY:
The aims of this study were to evaluate the pharmacokinetic properties and bioequivalence of two rebamipide preparations in healthy Korean male volunteers for generic substitution and to evaluate the association between the genetic polymorphisms in ABCB1 gene (exon 21 and 26) and rebamipide disposition.

DETAILED DESCRIPTION:
A randomized, single-dose, 2-period crossover design with a 7-day washout period was conducted in 30 healthy Korean male volunteers. Subjects were randomly assigned to receive a single 100-mg dose of the test or reference preparation of rebamipide, administered with 240 mL of water after a 12-hour overnight fast. All subjects were selected after passing a clinical screening procedure that included a physical examination and laboratory tests. Serum concentrations of rebamipide up to 12 hours after administration were determined using a validated HPLC method with fluorescence detection. Adverse events (AEs) were continuously monitored by clinical staff via observation, personal interview, and vital signs (temperature, blood pressure, heart rate) during the study period. All adverse events were recorded on the clinical record form per subject up to 1 week after the study. Pharmacokinetic parameters were determined using a noncompartmental method. The preparations were considered bioequivalent if the log-transformed ratios of AUC0-t, AUC0-∞, and Cmax were within the predetermined bioequivalence range (ie, 80-125%), as set by the US Food and Drug Administration (FDA) and Korean legislation. In vitro dissolution profiles of both preparations were examined and the influence of genetic polymorphisms in ABCB1 gene (P-glycoprotein) on the pharmacokinetics of rebamipide was also investigated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were selected after passing a clinical screening procedure that included a physical examination and laboratory tests (blood analysis; hemoglobin, hematocrit, RBC, WBC, platelet, differential counting of WBC, total proteins, albumin, ALT, AST, alkaline phosphatase, total bilirubin, cholesterol, creatinine, blood urea nitrogen, and fasting glucose and urine analysis; specific gravity, color, pH, sugar, albumin, bilirubin, RBC, WBC and cast).

Exclusion Criteria:

* Subjects possibly sensitive to this type of preparation,
* Subjects who had a history of any hepatic illness,
* Subjects who had a history of any renal illness,
* Subjects who had a history of any respiratory illness,
* Subjects who had a history of any endocrine illness,
* Subjects who had a history of any cardiovascular system illness,
* Subjects who had taken alcohol within 4 weeks prior to the study,
* Subjects who had taken other preparations within 4 weeks prior to the study.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-03; Primary Completion 2008-04 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Serum concentration of rebamipide | Pre-dose (to serve as a control) and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, and 12 hours after oral administration of rebamipide tablet (100 mg)

SECONDARY OUTCOMES:
Genetic polymorphisms in ABCB1 gene (exon 21 and 26) | A 3-mL blood sample was taken from each subject who participated in our bioequivalence studies before administration of rebamipide.

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Bok Lee, Ph.D., Principal Investigator — Institute of Bioequivalence and Bridging Study, College of Pharmacy, CNU
Locations (1):
- Institute of Bioeqivalence and Bridging Study, College of Pharmacy, CNU, Gwangju, South Korea

REFERENCES:
- [Derived] Cho HY, Yoon H, Park GK, Lee YB. Pharmacokinetics and bioequivalence of two formulations of rebamipide 100-mg tablets: a randomized, single-dose, two-period, two-sequence crossover study in healthy Korean male volunteers. Clin Ther. 2009 Nov;31(11):2712-21. doi: 10.1016/j.clinthera.2009.11.010. PMID 20110013